Statistical Analysis Plan: I6T-MC-AMBZ

A Multicenter, Phase 3b, Open-Label, Single-Arm Study to Investigate Bowel Urgency and its Relationship with Other Outcome Measures in Adults with Moderately to Severely Active Ulcerative Colitis Treated with Mirikizumab

NCT05767021

Approval Date: 27-Nov-2024

# Statistical Analysis Plan

#### **Protocol Title:**

A Multicenter, Phase 3b, Open-Label, Single-Arm Study to Investigate Bowel Urgency and its Relationship with Other Outcome Measures in Adults with Moderately to Severely Active Ulcerative Colitis Treated with Mirikizumab

**Protocol Number:** I6T-MC-AMBZ

Compound Number: Mirikizumab (LY3074828)

#### **Short Title:**

A Study to Investigate Bowel Urgency in Adults with Moderately to Severely Active Ulcerative Colitis Treated with Mirikizumab

**Acronym:** LUCENT-URGE

**Sponsor Name:** Eli Lilly and Company

Legal Registered Address: Indianapolis, Indiana, USA 46285

**Regulatory Agency Identifier Number(s)** 

**Registry** ID

U.S. Food and Drug Administration IND: 125444

European Medicines Agency EU trial number: 2022-502393-16-00

### **Confidential Information**

The information contained in this document is confidential and the information contained within it may not be reproduced or otherwise disseminated without the approval of Eli Lilly and Company or its subsidiaries

Note to Regulatory Authorities: This document may contain protected personal data and/or commercially confidential information exempt from public disclosure. Eli Lilly and Company requests consultation regarding release/redaction prior to any public release. In the United States, this document is subject to Freedom of Information Act (FOIA) Exemption 4 and may not be reproduced or otherwise disseminated without the written approval of Eli Lilly and Company or its subsidiaries.

Template Version: 1.0

# Statistical Analysis Plan Signature Page

Statistical Analysis Plan V3.0 (Dated 21NOV2024) for Protocol I6T-MC-AMBZ.

| | Name | Signature | Date (DDMMMYYYY) |
|---|---|---|---|
| Author: | PPD | Refer to eSignature | November 27, 2024 |
| Position: | Statistical Scientist | | |
| Company: | IQVIA | PPU | I approve this document<br>November 27, 2024 9:38:54 AM PS |

Upon review of this document, the undersigned approves this version of the Statistical Analysis Plan, authorizing that the content is acceptable for the reporting of this study.

| | Name | Signature | Date (DDMMMYYYY) |
|---|---|---|---|
| Approved By: | PPD | Refer to eSignature | November 22, 2024 |
| Position: | Statistical Scientist | | |
| Company: | IQVIA | PPD | I approve this document<br>November 22, 2024 6:56:20 AM JST |
| | | 519A7EFE2FBB4AE7 | 792F89CBC7A3D09A8 |
| Approved By: | PPD | Refer to eSignature | November 26, 2024 |
| Position: | Director-Statistics | | |
| Company: | Eli Lilly and Company | PPD | I approve this document |
| | | | November 26, 2024 12:33:08 F |

78AD8AAE33764642B15C7617F430CA4C

# **Table of Contents**

| Statist | ical Analysis Plan | 1 |
|---|---|---|
| Statist | ical Analysis Plan Signature Page | 2 |
| Table | of Contents | 3 |
| Abbre | viations and Definitions | 5 |
| Versio | n history | 9 |
| 1. | Introduction | 11 |
| 1.1. | Objectives, Endpoints, and Estimands | 11 |
| 1.2. | Study Design | |
| 2. | Statistical Hypotheses | 19 |
| 2.1. | Multiplicity Adjustment | 19 |
| 3. | Analysis Sets | 20 |
| 4. | Statistical Analyses | |
| 4.1. | General Considerations | |
| 4.1.1. | Analysis Methods | |
| 4.1.2. | Definition of Baseline | |
| 4.1.3. | Definition of Study Period Time Interval | |
| 4.1.4. | Missing Data Imputation | |
| 4.1.5. | Protocol Deviations | |
| 4.2. | Participant Dispositions, Baseline Characteristics and Medical History | |
| 4.2.1. | Demographics and Baseline Characteristics | |
| 4.2.2. | Non-UC Medical History | |
| 4.3. | Primary Endpoint Analysis | |
| 4.3.1. | Definition of Endpoint(s) | |
| 4.3.2. | Main Analytical Approach | |
| 4.4. | Secondary Endpoints Analysis | |
| 4.4.1. | Definition of Endpoint(s) | |
| 4.4.2.<br>4.5. | Main Analytical Approach | |
| CCI | Exploratory Endpoints Analysis | ∠0 |
| 4.6. | Safety Analyses | 27 |
| 4.6.1. | Extent of Exposure | 27 |
| 4.6.2. | Adverse Events | 27 |
| 4.6.3. | Clinical Laboratory Evaluations | 31 |
| 4.6.4. | Vital Signs and Other Physical Findings | 32 |
| 4.6.5. | Electrocardiograms | 32 |
| 4.6.6. | Immunogenicity | |
| 4.6.7. | Concomitant Therapy/ Procedure | |
| 4.6.8. | Substance Use | |
| 4.6.9. | Extraintestinal Manifestations of Inflammatory Bowel Disease | |
| 4.7. | Other Analyses | |
| 4.7.1. | Other variables and parameters | |
| 4.7.2. | Subgroup analyses | 33 |
| 4.8 Int | erim Analyses | 33 |

| 4.9 Cr | nanges to Protocol-Planned Analyses | 33 |
|--------|---------------------------------------------------------------|----|
| 5. San | nple Size Determination | 34 |
| 6. | Supporting Documentation | 35 |
| 6.1. | Appendix 1: Description and Derivation of Efficacy and Health | |
| | Outcome Endpoints | 35 |
| 6.2. | Appendix 2: Description of Analyses | 48 |
| 6.3. | Appendix 3: Demographic and Baseline Characteristics | |
| 6.4. | Appendix 4: Treatment Compliance | 56 |
| 6.5. | Appendix 5: Clinical Trial Registry Analyses | |
| 6.6. | Appendix 6: Study Visit or Week Definition for Daily Diary | |
| 7. | References | 60 |

# **Abbreviations and Definitions**

| Term | Definition |
|---|---|
| 5-ASA | 5-aminosalicylic acid |
| ADA | anti-drug antibody |
| AE | adverse event |
| AESI | adverse event of special interest |
| ALP | alkaline phosphatase |
| ALT | alanine aminotransferase |
| ANCOVA | analysis of covariance |
| AP | abdominal pain |
| APU | absorbent product use |
| AST | aspartate aminotransferase |
| ATC | anatomical therapeutic chemical |
| AZA | azathioprine |
| BMI | body mass index |
| BOCF | baseline observation carried forward |
| CCI | |
| CAP | continued access period |
| CFB | change from baseline |
| CI | confidence intervals |
| CMI | clinically meaningful improvement |
| CCI | |
| CSR | Clinical Study Report |
| ECG | electrocardiogram |
| eCRF | Electronic case report form; an electronic document designed to record all the protocol-required information to be reported to the sponsor for each trial participant |
| EIM | extraintestinal manifestation |
| ES | endoscopic subscore |
| FAS | Full Analysis Set |

| Term | Definition |
|---|---|
| CCI | |
| HLT | High Level Terms |
| IBD | Inflammatory Bowel Disease |
| CCI | |
| ICH | International Council for Harmonisation |
| informed consent | A process by which a participant voluntarily confirms their willingness to participate in a particular study, after having been informed of all aspects of the study that are relevant to the participant's decision to participate. Informed consent is documented by means of a written, signed, and dated informed consent form |
| interim analysis | An interim analysis is an analysis of clinical study data, separated into treatment groups, that is conducted before the final reporting database is created or locked |
| investigational product | A pharmaceutical form of an active ingredient or placebo being tested or used as a reference in a clinical trial, including products already on the market when used or assembled (formulated or packaged) in a way different from the authorized form, or marketed products used for an unauthorized indication, or marketed products used to gain further information about the authorized form. |
| ISR | Infusion/Injection Site Reactions |
| IV | intravenous |
| JAK | Janus Kinase |
| LLT | Lowest Level Term |
| MACE | major adverse cardiovascular events |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MI | multiple imputation |
| MMS | Modified Mayo Score |
| MMX | multi matrix colonic delivery technology |
| NAb | neutralizing anti-drug |
| NRI | nonresponder imputation |
| NRS | numeric rating scale |
| OI | opportunistic infections |

| Term | Definition |
|---|---|
| OR | odds ratio |
| Participant | Equivalent to CDISC term "subject": an individual who participates in a clinical trial, either as recipient of an investigational medicinal product or as a control |
| PD | Pharmacodynamics |
| PGA | Physician's Global Assessment |
| CCI | |
| | у |
| PK | pharmacokinetics |
| PT | preferred term |
| Q4W | once every 4 weeks |
| CCI | |
| QoL | quality of life |
| RB | rectal bleeding |
| CCI | |
| S1P | Sphingosine-1-phosphate |
| CCI | |
| SAE | serious adverse event |
| SAP | statistical analysis plan |
| SC | subcutaneous |
| Screen | The act of determining if an individual meets minimum requirements to become part of a pool of potential candidates for participation in a clinical study |
| CCI | |
| SF | stool frequency |
| SMD | standardized mean difference |
| SMQ | standardized MedDRA query |
| SoA | Schedule of Activities |
| SOC | system organ class |
| ТВ | tuberculosis |

# CONFIDENTIAL

| Term | Definition |
|---|---|
| TBL | total bilirubin level |
| TEAE | Treatment-emergent adverse event: An untoward medical occurrence that emerges during a defined treatment period, having been absent pretreatment, or worsens relative to the pretreatment state, and does not necessarily have to have a causal relationship with this treatment |
| TNF | tumor necrosis factor |
| UC | ulcerative colitis |
| ULN | upper limit of normal |
| UNRS | urgency numeric rating scale |
| CCI | |

# Version history

This Statistical Analysis Plan (SAP) for study I6T-MC-AMBZ is based on the protocol dated 16FEB2023.

 Table AMBZ.1.0.
 SAP Version History Summary

| SAP<br>Version | Approval<br>Date | Change | Rationale |
|---|---|---|---|
| 1.0 | 05APR2023 | Not Applicable | Original version |
| 2.0 | 24APR2024 | No Changes | Version updated to reflect yearly review |
| 3.0 | 21NOV2024 | Section 1.2 | Added details about the continued access period and continued access follow-up period start and stop details |
| | | Table AMBZ.4.1. | Updated language for period definition to accommodate Continued Access Period. |
| | | Section 4.3.2 Main analytical approach | Added explanation for odds ratio, Youden's index and standardized mean difference methods. |
| | | Table AMBZ4.2 | Switched binary and continuous variables in the ANCOVA analysis |
| | | Table AMBZ4.3 | Added footnotes to describe confidence interval analysis |
| | | Table AMBZ.4.3 Table AMBZ.6.2. | Updated APU for bowel urgency from bowel urgency measures to QoL measures, adjusted table for APU correlation analysis accordingly. |
| | | 4.6.2 Adverse Events | Added additional explanation for TEAE definition. Updated language that some safety analysis listings may be provided as appropriate. |
| | | 4.6.7 Concomitant<br>Therapy/ Procedure | Updated procedures from 'will be summarized' to 'may be summarized.' |
| | | Section 4.5.1 | Added CCI to analysis. |
| | | Table AMBZ.6.1. | Updated language for description and definition of |
| | | Table AMBZ.6.3 | Removed CCI from options on the prior therapy eCRF for biologic agents in footnote. |

# CONFIDENTIAL

| | Updated definition of location of disease |
|---|---|
| | Added a footnote for definition of S1P. |
| | Added prior advanced therapy exposure and prior advanced and biologic therapy failure. |
| | Updated prior therapy exposure and failure |
| Table AMBZ.6.4. | Updated language for daily diary time window calculation. |

## 1.

## Introduction

This document describes the rules and conventions to be used in presenting and analyzing the efficacy and safety data for the AMBZ study. It describes the data and details statistical analyses that will be performed.

There are no changes to the analyses described in the protocol.

# 1.1. Objectives, Endpoints, and Estimands

Table <u>AMBZ.1.1</u> shows the protocol-defined primary, secondary and exploratory objectives and endpoints of the study. The estimands (ICH E9R1 2017) associated with primary and secondary endpoint/analysis are also described in this section.

Table AMBZ.1.1. Study objectives and endpoints

| Objectives | Endpoints |
|---|---|
| Primary | |
| • To assess the improvement in bowel urgency severity at Week 12. | Change from baseline in bowel urgency severity (UNRS) score at Week 12. |
| Secondary | |
| <ul> <li>To assess the improvement in bowel urgency severity at Week .</li> <li>To assess the improvement in .</li> </ul> | |
| • To assess the improvement in CCI | |
| • To assess the proportion of participants achieving clinical remission and a UNRS score | |







Abbreviations: QoL = quality of life; UC = ulcerative colitis; UNRS = urgency numeric rating scale.







# 1.2. Study Design

This is a multicenter, open-label, single-arm Phase 3b study to investigate bowel urgency and its relationship with other outcome measures in participants with moderately to severely active UC treated with mirikizumab over a colored week period.

#### **Design**

The study will have 4 study periods:

## Period I ( days)

Participants must complete all Visit 1 screening activities within days prior to Visit 2. The screening endoscopy must occur within days prior to Visit 2.

| Period II ( weeks) |
|--------------------------------------------------|
| Participants will receive CCI mg mirikizumab CCI |
| Period III ( weeks) |
| Participants will receive CCI mg mirikizumab CCI |

Note: Participants planning to participate in continued access must complete self-administration training during at least 2 visits between Visits 6 and 9 (see Section 6.1.1 of protocol). Upon completion of all Visit 10 activities, eligible participants may enter the Continued Access Period.

#### Period IV

Participants who meet the following criteria should enter posttreatment follow-up, including completion of Visit 801:



#### Continued Access Period (CAP)

Participants who successfully completed Visit 10 and are eligible to enter the CAP. Participants will enter the CAP on the same day that they complete Visit 10 and remain until they discontinue from treatment in the CAP portion of the study. The CAP period will begin at dose of Visit 501 minus 1 minute and end at treatment discontinuation visit.

#### Continued Access Follow-up Period

Participants who entered the CAP and then discontinued treatment will enter the CAP follow-up period. They exit the CAP follow-up period when they complete Visit 901.

See <u>Figure AMBZ.1</u> in this SAP for schema. The Schedule of Activities (SoA) is described in Section 1.3 of protocol.



#### CCI

<sup>a</sup> Participants who are eligible for continued access should move directly from Visit 10 to Visit 501, on the same day, if possible. Visit 801 should not be performed.

b Optional Continued Access Period is described in Section 10.12 of the protocol.

# 2. Statistical Hypotheses

The primary objective is to assess the improvement from baseline in UNRS in participants treated with mirikizumab at Week. No formal hypothesis testing will be performed on the primary endpoint.

# 2.1. Multiplicity Adjustment

Multiplicity control is not applicable for this study.

# 3. Analysis Sets

Analysis sets are defined in <u>Table AMBZ.3.1</u> along with the planned analysis for each set. For both analysis sets, participants will be analyzed according to their assigned treatment unless otherwise specified.

Table AMBZ.3.1. Analysis sets

| Population | Description |
|---|---|
| Full Analysis | <b>Definition:</b> All participants who are assigned to treatment and receive at least 1 |
| Set (FAS) | (partial or complete) dose of study treatment (regardless of whether the participant |
| | does not receive the correct treatment, or otherwise does not follow the protocol). |
| | Purpose: Used for efficacy and health outcomes analysis |
| Safety Analysis | <b>Definition:</b> All participants who are assigned to treatment and receive at least 1 |
| Set | (partial or complete) dose of study treatment (regardless of whether the participant |
| | does not receive the correct treatment, or otherwise does not follow the protocol). |
| | Purpose: Used for safety-related analysis |

## 4. Statistical Analyses

## 4.1. General Considerations

Statistical analysis of this study will be the responsibility of Eli Lilly and Company (hereafter Lilly) or its designee. The statistical analyses will be performed using SAS® Version 9.4 or higher. The version of the Medical Dictionary for Regulatory Activities (MedDRA®) will be 24.0 or higher.

Any change to the data analysis methods in the protocol will require an amendment only if it changes a principal feature of the protocol. Additional exploratory analyses of the data will be conducted as deemed appropriate. Not all displays and analyses described in this SAP will necessarily be included in the clinical study report (CSR). Not all displays will necessarily be created as a "static" display. Some displays may be incorporated as interactive display tools instead of or in addition to a static display.

## 4.1.1. Analysis Methods

When reported, descriptive statistics will include the number of participants; mean, standard deviation, median, minimum, first and third quartile, and maximum for continuous measures; frequency counts and percentages for categorical measures; and estimate and 95% confidence intervals (CI) for correlation coefficients.

#### 4.1.2. Definition of Baseline

For efficacy and health outcomes analysis, baseline refers to the values or observations collected prior to or on the day of the initiation of study treatment in Study AMBZ, unless otherwise specified.

The baseline for variables collected as part of the daily diary (including the patient-reported outcomes components of the Modified Mayo Score, stool frequency (SF) and rectal bleeding (RB) subscores) will be calculated from valid daily diary entries obtained prior to baseline endoscopy preparation (see <a href="Appendix 6">Appendix 6</a>). The baseline endoscopy component of the Mayo Score will use the endoscopic appearance of the mucosa at the AMBZ screening endoscopy. For other efficacy and health outcome assessments, baseline is defined as the last non-missing assessment recorded on or prior to the date of the first study drug administration at Visit 2 (Week 0) in Study AMBZ.

Baseline for safety analysis is described in the Section 4.6.2 and Section 4.6.3.

Change from baseline will be calculated as the visit value of interest minus the baseline value. If a baseline value or the value at the visit is missing for a particular variable, then the change from baseline is defined as missing.

#### 4.1.3. Definition of Study Period Time Interval

<u>Table AMBZ.4.1</u> displays a list of study periods along with the definition of which participants will be considered to have entered the study period and when the individuals start and end the study period (refer to <u>Appendix 6</u> for additional details on study visits and study weeks). See Section 10.12 of protocol for more details about Continued Access Period (CAP).

To calculate the length of any time interval or time period in this study the following formula will be used:

 $Length\ of\ interval\ (days) = End\ Date\ -\ Interval\ Start\ Date\ +\ 1$ 

To convert any time length from days to years, the following formula will be used:

Length of interval (years) = Length of interval (days)/365.25

To convert any time length from days to weeks, the following formula will be used:

Length of interval (weeks) = Length of interval (days) /7

Only for the purpose of calculating the length of study period time intervals, the words "prior to" in <u>Table AMBZ.4.1</u> should be understood to mean "the day/time before" while the words "after" should be understood to mean "the day/time after." For the purpose of determining whether a date/time lies within an interval, these words are intended to convey whether the start or end of the period is inclusive of the specified date.

Table AMBZ.4.1. Definition of Main Study Period Time Intervals (excluding Continued Access Period)

| Main Study Period | <b>Interval Start Definition</b> | Interval End Definition |
|---|---|---|
| Period I (Screening): | Informed consent date | Prior to the start of study |
| All participants who sign | | treatment. |
| informed consent are considered | | |
| as entering the Screening Period. | | |
| Period II (CCI mg mirikizumab | At the date/time of first | Prior to first administration of |
| <u>cci</u> ): | administration of CCI mg | cci mg mirikizumab cci, or |
| All participants who received any | mirikizumab 🚾 | discontinuation of study |
| amount of mirikizumab are | | treatment, whichever is earlier |
| considered as entering Period II | | |
| and the treatment period. | | |
| Period III (CCI mg | At the date/time of first | Week Visit, or |
| mirikizumab <mark>COI</mark> ): | administration of CCI mg | discontinuation of study |
| All participants who received any | mirikizumab CCI | treatment, whichever is earlier |
| amount of mirikizumab on are | | |
| considered as entering Period III. | | |
| Period IV (Follow up) | After last date of any study | The maximum of the last |
| All participants who discontinued | treatment period for patients | study visit and study |
| mirikizumab treatment prior to | who did not enter CAP. | disposition date for patients |
| Visit 10, or completed Visit 10 | | who did not enter CAP. |
| and who did not enter CAP are | | |
| considered to have entered the | | |
| follow-up period. | | |

Abbreviations: CCI CAP = continued access period.

The CCI

The coweek analysis will include analysis through Week (Period III) but will not include analysis during the CAP. All safety and efficacy data will be included unless otherwise specified.

The CAP analysis will include a basic safety analysis, including disposition, analysis of AEs, vital signs, and lab data. Additional analysis during CAP will be performed as appropriate. All data from screening to end of CAP will be generally included.

#### 4.1.4. Missing Data Imputation

CCI



### 4.1.5. Protocol Deviations

Protocol deviations will be identified throughout the study. The protocol deviation categories will be described per Protocol Deviation Management Plan and Trial Issues Management Plan by clinical team. Important protocol deviations are defined in Protocol Deviation Management Plan as those deviations from the protocol that may significantly impact the completeness, accuracy and/or reliability of study data or that may significantly affect a subject's rights, safety or well-being.

# 4.2. Participant Dispositions, Baseline Characteristics and Medical History

The treatment disposition and study disposition will be summarized for the FAS population. The reason for discontinuation from treatment and from study will be included.

All FAS participants who discontinued from the study and/or study treatment during any period of the study will be listed with the reported study treatment discontinuation and study discontinuation times. If known, a reason for their discontinuation will be given.

## 4.2.1. Demographics and Baseline Characteristics

Summaries and listings of the demographic and baseline characteristics detailed in <u>Appendix 3</u> will be presented.

## **4.2.2.** Non-UC Medical History

Non-UC medical history will be collected on the Pre-Existing Conditions and Medical History case report form (CRF) and coded using MedDRA version 24.0 or higher. The version used to code medical history will be displayed in the outputs. All medical history will be summarized for the Safety Set by system organ class and preferred term. Prespecified medical history of liver and concurrent disease, hypersensitivity event, and associated person medical history of liver disease collected on the respective CRFs will also be summarized.

## 4.3. Primary Endpoint Analysis

#### 4.3.1. **Definition of Endpoint(s)**

The primary endpoint is defined in <u>Table AMBZ.1.1</u>, description and derivation of endpoints are described in <u>Table AMBZ.6.1</u>.

## 4.3.2. Main Analytical Approach

Analysis of the primary endpoint is described in Table AMBZ.6.2.

| The UNRS score at each time point of interest (baseline and Week ) will be summarized as a continuous measure for each participant as the average daily diary score over a day period. The difference between the UNRS score at Week and at baseline will be calculated for each participan |
|---|
| and averaged. <mark>CCI</mark> |
| CCI |

# 4.4. Secondary Endpoints Analysis

Section 4.1.4.

#### 4.4.1. **Definition of Endpoint(s)**

The secondary endpoint is defined in <u>Table AMBZ.1.1</u> Derivation details are described in <u>Table AMBZ.6.1</u>.

### 4.4.2. Main Analytical Approach

The analysis of the secondary endpoints is described in <u>Table AMBZ.6.2</u>. Descriptive summaries and CI will be provided for continuous and binary secondary endpoints as indicated in Section 4.1.1.

Analysis of association between secondary endpoints is described in <u>Table AMBZ.4.2</u> and <u>Table AMBZ.4.3</u>. At Week or Week these analyses will be performed among participants with available data that do not discontinue prior to the time point of interest.

**Table AMBZ.4.2.** Type of Endpoints and Association Analyses

| <b>Dependent Outcome</b> | <b>Explanatory Outcome</b> | Analysis |
|--------------------------|----------------------------|------------|
| Continuous | Continuous | |
| Continuous | Binary | <b>UUI</b> |
| Binary | Binary | |

Abbreviations: COl Youden's index (Youden 1950) (Kadel 2012); YI =

Table AMBZ.4.3. Type of Assessments and Endpoints for Association Analyses

| Assessments | <b>Endpoint Type</b> | Endpoint |
|---|---|---|
| Bowel Urgency | Continuous | UNRS, BUF, SDT, CCI |
| Assessments | | |
| | Binary | UNRS CMI, UNRS Remission |
| QoL/Function Measures | Continuous | CCI |
| | Binary | CCI |
| Symptom/ Symptom<br>Severity of UC | Continuous | CCI |
| | Binary | CCI |
| Histological Features | Continuous | (Analysis value, and CFB if applicable) |

| Assessments | <b>Endpoint Type</b> | Endpoint |
|------------------------------------|----------------------|----------|
| | Binary | |
| Additional Exploratory<br>Measures | Continuous | |



The odds ratio (OR) is calculated using logistic regression with 95% Wald confidence intervals, as implemented in SAS PROC LOGISTIC.

The Youden's Index (YI) and corresponding 95% confidence intervals are calculated using the equations presented in Youden, W.J. (1950).

The standardized mean difference (SMD) is calculated by mean difference divided by pooled standard deviation, where pooled standard deviation is obtained by taking the square root of the weighted average of the variances of each group in binary outcome, where the weights are the degrees of freedom of each group.

# 4.5. Exploratory Endpoints Analysis

Analysis of the exploratory endpoints other than gene expression endpoints are described in <u>Table AMBZ.6.2</u>. Analysis of associations between exploratory endpoints is described in <u>Table AMBZ.4.2</u> and AMBZ.4.3.





## 4.6. Safety Analyses

Safety will be assessed by describing the following: AEs, laboratory analytes, vital signs, and adverse events of special interest (AESIs). Additional analysis will be included if applicable.

#### 4.6.1. Extent of Exposure

Duration of exposure to study treatment will be summarized for the safety population. For the study periods of interest, exposure will be calculated as the time period length in years (see Section 4.1.3) with start and end dates described in Table AMBZ.4.1.

Total participant-years of exposure will be reported by treatment. Descriptive statistics will be provided for participant-weeks of exposure and the frequency of participants falling into different exposure ranges will be summarized. Exposure ranges will generally be reported in weeks using the following as a guide:

- >0 to <4 weeks,  $\ge 4$  weeks to <8 weeks,  $\ge 8$  weeks to <12 weeks,  $\ge 12$  weeks to <16 weeks,  $\ge 16$  weeks to <20 weeks,  $\ge 20$  weeks to <24 weeks,  $\ge 24$  weeks to <28 weeks.
- $>0, \ge 4$  weeks,  $\ge 8$  weeks,  $\ge 12$  weeks,  $\ge 16$  weeks,  $\ge 20$  weeks,  $\ge 24$  weeks,  $\ge 28$  weeks.

Additional exposure ranges may be considered if necessary.

Treatment compliance will be summarized as described in <u>Appendix 4</u>. Interruption of study treatment and the reasons drug not administered will be summarized for injection and infusion separately.

#### 4.6.2. Adverse Events

A treatment-emergent adverse event (TEAE) is defined as an event that first occurred or worsened in severity after baseline. Pre-existing events will be considered to determine TEAE. The MedDRA Lowest Level Term (LLT) will be used in the Treatment-emergent computation. The maximum severity for each LLT during the baseline period will be used as baseline. The treatment period will be included as postbaseline for the analysis. For events with a missing severity during the baseline period, it will be treated as 'mild' in severity for determining treatment-emergence. Events with a missing severity during the postbaseline period will be treated as 'severe' and treatment-emergence will be determined by comparing to baseline severity. For events occurring on the day of first taking study medication, the start times of the study treatment and AE will be used to determine whether the event was pre-versus posttreatment. If start time for the AE is missing, it will be assumed to have started in the postbaseline period.

In an overview table, the number and percentage of participants with at least 1 TEAE, serious adverse event (SAE), fatal SAE, or discontinuation from study treatment due to an AE will be summarized. TEAEs (all and by maximum severity), SAEs, including deaths, and AEs that lead to treatment discontinuation will be summarized and analyzed by MedDRA system organ class (SOC) and PT or by PT alone. Potential AESIs will be summarized, which include:



See <u>Section 4.6.2.1</u> for detailed description on AESI.

Summary tables as described in <u>Table AMBZ.4.4</u> will be presented. Summary tables will include the number and percentage of participants reporting an event. For events that are gender-specific (as defined by MedDRA), the number of participants at risk will include only participants from the given gender. Listing of AEs may be provided as deemed appropriate.

## **Table AMBZ.4.4.** Summary Tables Related to Adverse Events

| Analysis |
|---|
| Overview of AEs |
| Summary of TEAE PTs by decreasing frequency |
| Summary of TEAE PTs occurring in >=1% of participants by decreasing frequency |
| Summary of TEAE PTs by decreasing frequency within SOC |
| Summary of TEAE PTs by maximum severity by decreasing frequency within SOC |
| Summary of SAE PTs by decreasing frequency within SOC |
| Summary of fatal SAE PTs by decreasing frequency within SOC |
| Summary of AEs leading to study treatment discontinuation by decreasing frequency of PTs within SOC |
| Listing of SAEs |

Abbreviations: AE = adverse event; AESI = adverse event of special interest; PT = preferred term; SAE = serious adverse event; SOC = system organ class; TEAE = treatment-emergent adverse event.

## 4.6.2.1. Special Safety Topics including Adverse Events of Special Interest

This section includes areas of interest whether due to observed safety findings, potential findings based on drug class, or safety topics anticipated to be requested by a regulatory agency for any reason. In general, potential AESIs relevant to these special safety topics will be identified by one or more standardized MedDRA query(ies) (SMQs), by a Lilly defined MedDRA PT listing based upon the review of the most current MedDRA Version, or by TE relevant laboratory changes, as described below. Additional special safety topics may be added as warranted.

Unless otherwise specified, the treatment-emergent AESIs will be summarized for the safety population.

Full details of the search terms and rules for deriving AESIs in each of the sections below are described in the compound level safety standards along with information about the types of summaries and listings to be provided.







## 4.6.3. Clinical Laboratory Evaluations

As described more fully in compound level safety standards and in the laboratory-related PhUSE white papers [PhUSE 2013; PhUSE 2015], the clinical laboratory evaluations will be summarized with the following displays described in <u>Table AMBZ.4.5</u>:

## Table AMBZ.4.5. Summaries/Displays/Analysis for Clinical Laboratory Evaluations

#### **Analysis**

Box plots of observed values (and change from baseline values) by visit. Change from baseline to last observation will be summarized within the box plot of changes (rightmost column), and descriptive summary statistics will be included in a table below the box plot.

Treatment-emergent abnormal high lab values (i.e., participants shifting from a normal/low maximum baseline value to a high maximum postbaseline.

Scatter plot of maximum (minimum) postbaseline value vs. maximum (minimum) baseline value if appropriate.

Shift tables showing the number of participants who shift from each category of maximum (minimum) baseline observation to each category of maximum (minimum) postbaseline observation. Here categories may be low, normal or high with cutoffs defined in the compound level safety standards.

For these displays, the postbaseline periods will be identical to those described in <u>Table AMBZ.4.1</u>. Postbaseline measurement for continuous analysis (e.g., boxplots) will include *only* 

scheduled measurements, while postbaseline categorical analysis (e.g., shifts) will include *both* scheduled and unscheduled measurements.

For any lab performed on the day of first taking study medication at the start of the postbaseline period, the start time of the study treatment will be used to determine whether the lab was preversus postbaseline. If time for the lab is missing, it will be assumed to be in the baseline period (i.e., we assume the protocol-defined order of procedures was followed). Following the compound level safety standards, for some labs a safety concern may exist for only high (or only low) values. For these labs, displays with only maximum (or minimum) values will be used, and shift tables will be presented accordingly.

Hepatic serology, hematology, chemistry and coagulation tests will be done by local laboratory. Descriptive statistics of the test results will be summarized in a table. Summary will be done using standardized units (SI).

Screening assessment of Tuberculosis (TB) and evaluation of TB during the study will be listed, as appropriate.

### 4.6.4. Vital Signs and Other Physical Findings

As described more fully in compound level safety standards and in the vital signs-related PhUSE white papers [PhUSE 2013; PhUSE 2015], vital signs will be summarized similarly to the clinical laboratory evaluation (see Section 4.6.3). For vital signs, the low and high limits are based on a combination of a specified value and a change or percentage change. In this case, the PhUSE white paper recommends providing scatter plots and shifts to low/high. Boxplots will also be presented.

## 4.6.5. Electrocardiograms

Complete electrocardiogram (ECG) data will not be part of the clinical database for this study. Any clinically significant findings from ECGs that result in a diagnosis and that occur after the participant receives the first dose of the investigational treatment will be reported to Lilly or its designee as an AE via eCRF. Aside from standard AE summary tables no additional analysis of ECG data will be performed.

#### 4.6.6. Immunogenicity



Compound level safety standards will be followed in the analyses of immunogenicity. Listings of immunogenicity assessments may be provided along with the summary of specified TEAEs by TE ADA status. The summary of TE ADA and NAb status may be produced as appropriate. Additional assessments of the relationship between immunogenicity and efficacy will be performed as deemed appropriate.

#### 4.6.7. Concomitant Therapy/ Procedure

Medications will be classified into anatomical therapeutic chemical (ATC) drug classes using the latest version of the World Health Organization (WHO) drug dictionary. Medication start and stop

dates will be compared to the date of first dose of treatment to allow medications to be classified as Concomitant for treatment period.

Prior medications are those medications that start and stop prior to the date of first dose of study treatment. Concomitant medications are those medications that start before, on or after the first dose of study treatment and end on or after the date of first dose of study treatment or are ongoing at the end of the study. If it cannot be determined whether a medication is concomitant or not due to a partial or missing date, the medication will be treated as concomitant.

Concomitant medications may be summarized by ATC and preferred term for the Safety Set and sorted by descending frequency. Prespecified concomitant therapy of acetaminophen/paracetamol may also be summarized.

Concomitant UC-related surgeries will be summarized by procedure type for the Safety Set, as needed. The other procedures including hepatic monitoring procedures and endoscopic procedures will be listed.

Prior and concomitant use of vaccines may be listed as appropriate.

#### 4.6.8. Substance Use

Substance use of alcohol, caffeine, tobacco, nicotine, and recreational drug at screening and change in substance use by visit may be listed, as appropriate.

## 4.6.9. Extraintestinal Manifestations of Inflammatory Bowel Disease

Extraintestinal manifestations (EIM) of inflammatory bowel disease will be reported in the Inflammatory Bowel Disease (IBD) EIM eCRF by visit and will be summarized by prespecified term.

## 4.7. Other Analyses

Reference the analyses described in Appendix 5 in this section.

## 4.7.1. Other variables and parameters

The pharmacokinetic/pharmacodynamics (PK/PD) analyses will be conducted by the PK/PD and Pharmacometrics group at Eli Lilly.

#### 4.7.2. Subgroup analyses

Subgroup analyses may be conducted for all primary and secondary endpoints in the FAS population. The subgroups to be analyzed are listed in <u>Table AMBZ.6.3</u>.

# 4.8 Interim Analyses

CCI

# **4.9 Changes to Protocol-Planned Analyses**

There are no changes to the analyses described in the protocol.

## 5. Sample Size Determination

Approximately 160 participants will be assigned to study intervention. The sample size was determined by considering the precision of the estimated correlation between endpoints. Simulations were performed for both binary and continuous measures where the true correlation varied between CCI . The average half width of the 95% CI for the correlations at Week varied between under considered assumptions for an overall sample size of 160. The average half width of the 95% CI varied between for endpoints during the maintenance period under the assumption that CCI of participants could discontinue early from the study.

Additionally, the proposed sample size of 160 participants is considered sufficient to have power to detect a significant (non-zero) change from baseline in UNRS at Week (primary endpoint).

# **6.** Supporting Documentation

# **6.1.** Appendix 1: Description and Derivation of Efficacy and Health Outcome Endpoints

All binary endpoints will be coded as Yes/No, unless otherwise specified.

Table AMBZ.6.1. Description and Derivation of Efficacy, Safety and Health Outcomes Measures and Endpoints

| Measure | Description | Variable | Derivation / Comment | Definition of<br>Missing |
|---|---|---|---|---|
| Mayo Score and components | The Mayo score is a composite instrument to measure Ulcerative Colitis disease activity. It is comprised of the following 4 subscores: | SF subscore | | |
| | | RB subscore | | |
| | | ES subscore | | |
| Measure | Description | Variable | Derivation / Comment | Definition of<br>Missing |
|---|---|---|---|---|
| | CCI | PGA subscore | | |
| | | Clinical Remission | | |
| | | Alternate Clinical<br>Remission | | |
| | | Modified Mayo Score | _ | |
| | | (MMS) | | |
| | | Clinical Response | | |
| | | Symptomatic Remission | _ | |
| | | Symptomatic Remission | | |
| | | SF component of | _ | |
| | | clinical remission RB component of | _ | |
| | | clinical remission | | |

| Measure | Description | Variable | Derivation / Comment | Definition of<br>Missing |
|---|---|---|---|---|
| | | Endoscopic<br>Normalization Absolute SF | | |
| | | Endoscopic<br>Remission | | |
| Urgency NRS | The Urgency numeric rating scale (NRS) is a single item that measures the severity for the urgency (sudden or immediate need) to have a bowel movement in the past 24 hours using | Urgency NRS | | |
| | an 11-point NRS ranging from 0 ("no urgency") to 10 ("worst possible urgency"). | Change from Baseline<br>Urgency NRS | | |
| | | Urgency NRS CMI (>=3 Point Improvement) | | |
| | | Alternate Urgency NRS<br>Remission | | |
| | | Urgency NRS Remission | | |







| Measure | Description | Variable | Derivation / Comment | Definition of<br>Missing |
|---|---|---|---|---|
| | | Normal Number of Stools | Use the single item collected | CCI |
| | | CCI | Use the single item collected | - |
| | | CCI | CCI | |
| | | CCI | CCI | |













# **6.2.** Appendix 2: Description of Analyses

 Table AMBZ.6.2.
 Description of Efficacy/Health Outcomes Analyses

| Measure | Variable | Analysis Method | Population | Time Point(s) |
|---|---|---|---|---|
| Urgency NRS | CFB in Urgency<br>NRS Score (Primary<br>Endpoint) | Descriptive summaries, including 95% CI | FAS | Baseline (if applicable), CCI |
| | UNRS CMI | Descriptive summaries, including 95% CI | | |
| | UNRS Remission | Descriptive summaries, including 95% CI | | |
| | Alternate UNRS<br>Remission | Descriptive summaries, including 95% CI | | |
| CCI | CCI | Descriptive summaries, including 95% CI | | |
| | CCI | Descriptive summaries, including 95% CI | | |
| CCI | CCI | Descriptive summaries, including 95% CI | | |
| | CCI | Descriptive summaries, including 95% CI | | |
| CCI | CCI | Descriptive summaries, including 95% CI | | |
| | CCI | Descriptive summaries, including 95% CI | | |
| Mayo Score<br>and Urgency<br>NRS | Clinical Remission and Urgency NRS | Descriptive summaries, including 95% CI | | |
| | Clinical Response<br>and Urgency NRS<br>point<br>Improvement | Descriptive summaries, including 95% CI | | |
| Bowel Urgency | | | • | - |
| Urgency NRS | UNRS | coefficient with CCI | FAS | Baseline (if applicable), CCI |
| | CFB UNRS | coefficient with CFB CCI | | |
| | UNRS CMI, UNRS<br>Remission | ANCOVA with column and CFB column | | |
| CCI | CCI | coefficient with CCI | | |
| | CCI | coefficient with CFB CCI | | |
| QoL Analysis | <u> </u> | | | |
| CCI | CCI | Descriptive summaries, including 95% CI | FAS | Baseline (if applicable), CCI |
| | CCI | Descriptive summaries, | 7 | |

| Measure | Variable | Analysis Method | Population | Time Point(s) |
|---|---|---|---|---|
| | | including 95% CI | | |
| | | Descriptive summaries, including 95% CI | FAS | Baseline (if applicable), CCI |
| | | Descriptive summaries, | | applicable), cel |
| | | including 95% CI | | |
| | | Descriptive summaries, | | |
| | | including 95% CI | | |
| | | Descriptive summaries, including 95% CI | | |
| | | Descriptive summaries, | | |
| | | including 95% CI | | |
| Bowel | UNRS, CCI | CCI | | |
| Urgency<br>Analysis | | Score and component subscores | | |
| Allalysis | | CCI | | |
| | | component scores | | |
| | | ccl | | |
| | | Pearson + Spearman correlation | | |
| | | coefficient with APU | | |
| | CFB UNRS, CFB | CCI | | |
| | CFB | coefficient with CFB CCI and | | |
| | CCI | component scores | | |
| | | coefficient with CFB CCI | | |
| | | component scores | | |
| | | Pearson + Spearman correlation | | |
| | | coefficient with CFB CCI | | |
| | | coefficient with CFB APU | | |
| | | ANCOVA with CC | | |
| | | ANCOVA with CC | | |
| Bowel | UNRS CMI, UNRS<br>Remission | ANCOVA with CFB CCI and | | |
| Urgency<br>Analysis | Remission | ANCOVA with Column and | | |
| | | components score | | |
| | | ANCOVA with CC | | |
| | | components score | | |
| | | ANCOVA with CFB ccl components score | | |
| | | ANCOVA with CFB CC | | |
| | | ANCOVA with CC | | |
| | | ANCOVA with CFB CC | | |
| | | ANCOVA with CO | | |
| | | OR, YI with CCI remission OR, YI with CCI response | | |
| IIC Compton /C | symptom Severity Analy | | | |
| oc symptom/S | symptom Severity Analy | 7515 | | |
| CCI | CCI | Descriptive summaries, | FAS | Baseline (if |
| | | including 95% CI | | applicable), CCI |
| CCI | CCI | Descriptive summaries, | | |

| Measure | Variable | Analysis Method | Population | Time Point(s) |
|---|---|---|---|---|
| | | including 95% CI | | |
| Absolute SF | Absolute SF Score | Descriptive summaries, | | |
| 2.5 | ~~ . | including 95% CI | | |
| Mayo | SF subscore | Descriptive summaries, | | |
| | RB subscore | including 95% CI Descriptive summaries, | - | |
| | KD subscore | including 95% CI | | |
| | MMS | Descriptive summaries, | | |
| | | including 95% CI | | |
| | Symptomatic | Descriptive summaries, | | |
| | Remission | including 95% CI | | |
| | Clinical Remission | Descriptive summaries, | | |
| | City is all Decreases | including 95% CI | - | |
| | Clinical Response | Descriptive summaries, including 95% CI | | |
| | Alternate Clinical | Descriptive summaries, | - | |
| | Remission | including 95% CI | | |
| Mayo | Endoscopic | Descriptive summaries, | FAS | Baseline (if |
| | Normalization | including 95% CI | | applicable), CCI |
| | Endoscopic | Descriptive summaries, | | |
| E C NDC | Remission | including 95% CI | | |
| Fatigue NRS | Fatigue NRS Score | Descriptive summaries, including 95% CI | | |
| Abdominal | Abdominal Pain | Descriptive summaries, | - | |
| Pain NRS | NRS Score | including 95% CI | | |
| Nocturnal stool | | Descriptive summaries, | | |
| | Score | including 95% CI | | |
| CCI | CCI | Descriptive summaries, | | |
| | | including 95% CI | | |
| | CCI | Descriptive summaries, | | |
| | | including 95% CI | | |
| Bowel | UNRS, CCI | CCI | | |
| Urgency<br>Analysis | | coefficient with CCI | | |
| Allalysis | | coefficient with CCI | | |
| | | CCI | 1 | |
| | | coefficient with Mayo SF | | |
| | | CCI | | |
| | | coefficient with Absolute SF | | |
| | | CCI | | |
| | | coefficient with Mayo RB | - | |
| | | coefficient with AP NRS | | |
| | | CCI | 1 | |
| | | coefficient with Fatigue NRS | | |
| | | Pearson + Spearman correlation | | |
| | | coefficient with Nocturnal Stool | | |
| | | ANCOVA with clinical response | | |
| | | ANCOVA with endoscopic remission | - | |
| | | ANCOVA with endoscopic remission ANCOVA with endoscopic | - | |
| | | normalization | | |
| | | ANCOVA with symptomatic | 1 | |

| Measure | Variable | Analysis Method | Population | Time Point(s) |
|---|---|---|---|---|
| | | remission | | |
| | CED IDIDG CED | ANCOVA with CC | | |
| | CFB UNRS, CFB | coefficient with CFB CCI | | |
| | | coefficient with CFB Mayo SF | | |
| | | CCI | | |
| | | coefficient with CFB Absolute SF | | |
| | | coefficient with CFB Mayo RB | | |
| | | coefficient with CFB AP NRS | | |
| | | coefficient with CFB Fatigue NRS | | |
| | | CCI | | |
| | | coefficient with CFB Nocturnal Stool ANCOVA with clinical response | | |
| | | ANCOVA with clinical remission | | |
| | | ANCOVA with endoscopic remission | | |
| | | ANCOVA with endoscopic | | |
| | | normalization ANCOVA with symptomatic | | |
| | | remission | | |
| Bowel | CFB UNRS, CFB | ANCOVA with CC | FAS | Baseline (if |
| Urgency | cci , CFBcci | | | applicable), CCI |
| Analysis | | | | |
| | UNRS CMI, UNRS | ANCOVA with CFB CC | | |
| | Remission | ANCOVA with CFB Mayo SF | | |
| | | ANCOVA with CFB Absolute SF | | |
| | | ANCOVA with CFB Mayo RB | | |
| | | ANCOVA with CFB AP NRS | | |
| | | ANCOVA with CFB Fatigue NRS | | |
| | | ANCOVA with CFB Nocturnal Stool | | |
| | | OR, YI with clinical response OR, YI with clinical remission | | |
| | | OR, YI with endoscopic remission | | |
| | | OR, YI with endoscopic | | |
| | | normalization | | |
| | | OR, YI with symptomatic remission | | |
| | | OR, YI with Bristol Loose Stool | | |
| Exploratory Ana | alyses | Description annual control 100 | | Dogalina (:f |
| | | Descriptive summaries, including 95%CI | FAS | Baseline (if applicable), CCI |
| | | Descriptive summaries, including 95% CI | | |
| | | Descriptive summaries, including | | |
| | | | | • |

| Measure | Variable | Analysis Method | Population | Time Point(s) |
|---|---|---|---|---|
| | | 95% CI | | (-) |
| | | Descriptive summaries, including 95% CI | | |
| Bowel<br>Urgency | UNRS, CCI | coefficient with CCI | | |
| Analysis | | coefficient with CCI | | |
| | | coefficient with WIS | _ | |
| | | coefficient with SAA | | |
| | | ANCOVA with CCI | | |
| Bowel | UNRS, CCI | ANCOVA with CCI | FAS | Baseline (if |
| Urgency<br>Analysis | | ANCOVA with CCI | | applicable), CCI |
| | | ANCOVA with CCI | | |
| | | ANCOVA with CCI | | |
| | | AIVEOVA WILLI | | |
| | | ANCOVA with CCI | | |
| | | coefficient with CCI | | |
| | | coefficient with CCI | | |
| | CFB UNRS, CFB | coefficient with CFB CCI | | |
| | | coefficient with CFB CCI | | |
| | | CCI coefficient with CCI | | |
| | | coefficient with CCI CFB | | |
| | UNRS CMI, UNRS<br>Remission | OR, YI with CCI | | |
| | Kemission | OR, YI with CC | _ | |
| | | OR, YI with CCI | _ | |
| | | , 11 mm | | |

| Measure | Variable | Analysis Method | Population | Time Point(s) |
|---------|----------------|---------------------|------------|---------------|
| | | OR, YI with CCI | | |
| | | OR, YI with CCI | | |
| | | OR, YI with CCI | | |
| | UNRS CMI, UNRS | ANCOVACCI | | |
| | Remission, | ANCOVA with CCI CFB | | |
| | | ANCOVA with CC | | |
| | | ANCOVA with CC CFB | | |



Additional exploratory analysis will be performed as appropriate.

## **6.3.** Appendix 3: Demographic and Baseline Characteristics

Participant demographic variables and baseline characteristics will be summarized for the FAS. The baseline characteristics of participants entering additional study periods may also be summarized if necessary. The continuous variables will be summarized using descriptive statistics and the categorical variables will be summarized using frequency counts and percentages. No inferential analysis for the comparability of baseline covariates across treatment groups will be performed. By-participant listings of basic demographic characteristics (i.e., gender, age, body weight, race, ethnicity, geographic region, prior biologic/ Janus Kinase (JAK)/ Sphingosine-1-phosphate (S1P) use and/or failure, corticosteroid use at baseline, duration of disease, and disease location) for the FAS will be provided as deemed appropriate.

<u>Table AMBZ.6.3</u> describes the specific variables and how they will be summarized. The final column specifies variables used for the efficacy subgroup analysis.

Table AMBZ.6.3. Participant Characteristics (and Variables for Subgroup Analysis)

| Variable | Continuous<br>Summary | Categorical Summary | Subgroup<br>Analysis <sup>a</sup> |
|---|---|---|---|
| Demographic Characteristics | | | |
| Age <sup>b</sup> | Yes | <65 years, ≥65 years | |
| Age | res | <40 years, ≥40 years | |
| Sex | No | Male, Female | |
| | | Male <40 years, Male ≥40 years, Female | |
| Age within Sex | No | <40 years, Female ≥40 years | |
| Ethnicity | No | Hispanic/Latino, Non-Hispanic/Non-Latino | |
| | | American Indian/Alaska Native, Asian, | |
| Race | No | Black/African American, Native Hawaiian | |
| | | or other Pacific Islander, White, or Multiple | |

| Variable | Continuous<br>Summary | Categorical Summary | Subgroup<br>Analysis <sup>a</sup> |
|---|---|---|---|
| | No | North America, Europe | - |
| Geographic Region | No | North America, East Europe, West Europe | X |
| II: 1// | No | By Country (listed in other documents) | |
| Height (cm) | Yes | None | |
| Weight (kg) | Yes | <80 kg, ≥80 kg<br><100 kg, ≥100 kg | |
| BMI <sup>c</sup> | Yes | Underweight ( $<18.5 \text{ kg/m2}$ ), Normal ( $\ge18.5 \text{ and } <25 \text{ kg/m2}$ ), Overweight ( $\ge25 \text{ and } <30 \text{ kg/m2}$ ), Obese ( $\ge30 \text{ and } <40 \text{ kg/m2}$ ), Extreme obese ( $\ge40 \text{ kg/m2}$ ) | |
| Prior UC Therapies | | | |
| Prior corticosteroid <sup>d</sup> failure <sup>e</sup> | No | Failed, Not failed | |
| Prior immunomodulator failure | No | Failed, Not failed | |
| Prior JAK inhibitorh exposure | No | Ever, Never | |
| Prior JAK inhibitor <sup>h</sup> failure <sup>e</sup> | No | Failed, Not failed | |
| Prior biologic agents exposure | No | Ever, Never | |
| Prior biologic agents failure | No | Failed, Not failed | |
| Number of prior biologic agents <sup>g</sup> used | No | 0, 1, 2, 3, >3 | |
| Number of failed <sup>e</sup> biologic agents <sup>g</sup> | No | 0, 1, 2, 3, >3 | |
| Number of prior JAK inhibitor <sup>h</sup> used | No | 0, 1, 2 | |
| Number of failed <sup>e</sup> JAK inhibitor <sup>h</sup> | No | 0, 1, 2 | |
| Prior advanced <sup>i</sup> therapy exposure | No | Ever, Never | |
| Prior advanced <sup>i</sup> therapy failure | No | Failed, Not failed | X |
| Number of prior advanced i therapy used | No | 0, 1, 2, 3, >3 | |
| Number of failed advanced i therapy | No | 0, 1, 2, 3, >3 | |
| Prior S1P therapy <sup>n</sup> exposure <sup>e</sup> | No | Ever, Never | |
| Prior S1P therapy <sup>n</sup> failure <sup>e</sup> | No | Failed, Not Failed | |
| Baseline UC Therapies Baseline Corticosteroid use <sup>j</sup> | No | Yes, No | v |
| Baseline Prednisone equivalent | Yes | None Yes, No | X |
| dose Baseline Budesonide MMX <sup>k</sup> | No | Yes, No | |
| Baseline Beclomethasone | No | Yes, No | |
| dipropionate Baseline Oral Aminosalicylates <sup>1</sup> dose | Yes | None | |
| Baseline immunomodulator use <sup>j</sup> | No | Yes, No | |
| Baseline Antidiarrheals/<br>Antispasmodics use | No | Yes, No | |
| Baseline Disease Characteristics | | | |
| Duration of UC <sup>m</sup> | Yes | <pre>&lt;1 year, ≥1 to &lt;3 years, ≥3 year to &lt;7 years,<br/>≥7 years</pre> | |
| Age at Diagnosis of UCb | Yes | $<6, \ge 6 \text{ to } < 10 \text{ year}, \ge 10 \text{ to } < 17 \text{ years}, \ge 17$ | |

| Variable | Continuous<br>Summary | Categorical Summary | Subgroup<br>Analysis <sup>a</sup> |
|---|---|---|---|
| | | year to <40 years, ≥40 years | - |
| Baseline Disease Location <sup>o</sup> | No | Ulcerative Proctitis, Left-sided UC (distal UC), Extensive UC (pancolitis) | X |
| Baseline Fecal Calprotectin | Yes | ≤250 μg/g, >250 μg/g | X |
| Baseline Modified Mayo Score | Yes | Mild (1-3), Moderate (4-6), Severe (7-9) | X |
| Baseline Total Mayo Score | Yes | Mild (3-5), Moderate (6-9), Severe (10-12) | |
| Baseline Endoscopic Mayo<br>Subscore | No | Possible values of 4-point scale in <u>Table</u> AMBZ.6.1 | X |
| Baseline Stool Frequency Mayo<br>Subscore | Yes | Possible values of 4-point scale in <u>Table</u> AMBZ.6.1 | |
| Baseline Absolute Value Stool<br>Frequency Mayo Subscore | Yes | Possible values of 4-point scale in <u>Table</u> AMBZ.6.1 | |
| Baseline Absolute Stool<br>Frequency | Yes | None | |
| Baseline Rectal Bleeding (RB) Mayo Subscore | Yes | Possible values of 4-point scale in <u>Table</u><br><u>AMBZ.6.1</u> | |
| Baseline IBDQ Total Score and<br>Domain Scores | Yes | None | |
| Baseline Urgency NRS | Yes | None | |
| Baseline Abdominal Pain NRS | Yes | <4,≥4 | |
| Baseline Patient's Global Rating of Severity (PGRS) | Yes | None | |
| Baseline Nocturnal Stool | Yes | Yes (≥1), No (0) | |
| Baseline Fatigue NRS | Yes | Yes (1-10), No (0) | |
| Baseline Bristol Stool Scale | Yes | Not Loose Stool $(1-5)$ , Loose Stool $(6-7)$ | |
| Baseline Stool Deferral Time | Yes | No | |
| Baseline Stool Deferral Time<br>Category | Yes | 0: ≥ 15 min<br>1: ≥ 5 to < 15 min<br>2: ≥ 2 to < 5 min<br>3: ≥ 1 to < 2 min<br>4: < 1 min | |
| Baseline Bowel Urgency<br>Frequency | Yes | None | |
| Other Baseline Patient-Reported | | | |
| Alcohol Use | No | Never, Current, Former | |
| Caffeine Use | No | Never, Current, Former | |
| Tobacco Use | No | Never, Current, Former | |
| Nicotine Use | No | Never, Current, Former | |
| Recreational Drug Use | No | Never, Current, Former | |

Abbreviation: 5-ASA = 5-aminosalicylic acid; 6-MP = 6-mercaptopurine; ATC= Anatomical Therapeutic Chemical; AZA = azathioprine; eCRF = electronic clinical report form; IBDQ = Inflammatory Bowel Disease Questionnaire; JAK = Janus Kinase; MMX = multi matrix colonic delivery technology; MTX = Methotrexate; NRS = numeric rating scale; PGA = Physician's Global Assessment; S1P = Sphingosine-1-phosphate; TB = tuberculosis; TNF = tumor necrosis factor; UC = ulcerative colitis.





## **6.4.** Appendix 4: Treatment Compliance

Treatment compliance with IP will be summarized for participants who enter the treatment period. The treatment compliance of patents while being treated during other study periods may also be summarized if necessary. Treatment compliance for each participant will be calculated as:

 $Treatment\ compliance\ (\%)$   $=100\times\frac{{\it Total\ number\ of\ study\ drug\ administration\ visits}}{{\it Total\ number\ of\ study\ drug\ administration\ visits\ planned\ per\ protocol}}$ 

The "Total number of study drug administration visits planned per protocol" is based on the administration number of planned visits before the participant discontinued study drug. Each participant will be defined as having had a study drug administration visit on a given date if:

- For visits where the participant is to receive an IV infusion, they received the planned dose (i.e.., a partial dose does not count) as derived from the Exposure eCRF page
- For visits where the participant is to receive SC injections, they received the planned number of injection doses (i.e., 2 doses) as derived from the Exposure eCRF page

"Overall compliance" with therapy is defined as having at least 80% treatment compliance. Proportions of participants who satisfy the definition of overall compliance during the treatment period will be summarized for FAS population.

## **6.5.** Appendix 5: Clinical Trial Registry Analyses

Additional analyses will be performed for the purpose of fulfilling the Clinical Trial Registry (CTR) requirements.

Analyses provided for the CTR requirements include the following:

• Summary of AEs, provided as a dataset which will be converted to an XML file. Both SAEs and 'Other' AEs are summarized: by MedDRA PT.

- An AE is considered 'Serious' whether or not it is a TEAE.
- An AE is considered in the 'Other' category if it is both a TEAE and is not serious. For each SAE and 'Other' AE, for each term, the following are provided:
  - o the number of participants at risk of an event
  - o the number of participants who experienced each event term
  - o the number of events experienced.
- Consistent with www.ClinicalTrials.gov requirements, 'Other' AEs that occur in fewer than 5% of participants/subjects may not be included if a 5% threshold is chosen (5% is the minimum threshold).
- AE reporting is consistent with other document disclosures, for example, the CSR, manuscripts, and so forth.

### **6.6.** Appendix 6: Study Visit or Week Definition for Daily Diary

Weekly summary measures of daily diary data will be created for each participant. The 7-day period associated with each week will be defined using a visit centric approach. The table below displays the interval for each week.







#### 7. References

Geboes K, Riddell R, Ost A, Jensfelt B, Persson T, Löfberg R. A reproducible grading scale for histological assessment of inflammation in ulcerative colitis. Gut. 2000 Sep;47(3):404-9. doi: 10.1136/gut.47.3.404. PMID: 10940279; PMCID: PMC1728046.

Guyatt G, Mitchell A, Irvine EJ, et al. A new measure of health status for clinical trials in inflammatory bowel disease. *Gastroenterology*. 1989;96(30):804-810. https://doi.org/10.1016/S0016-5085(89)80080-0

International Conference on Harmonization. ICH E9 (RI): Addendum to statistical principles for clinical trials on choosing appropriate estimands and defining sensitivity analyses in clinical trials.2017. Available at:

https://www.fda.gov/downloads/Drugs/GuidanceComplianceRegulatoryInformation/Guidances/UCM582738.pdf

Irvine EJ, Feagan B, Rochon J, et al. Quality of Life: a valid and reliable measure of therapeutic efficacy in the treatment of inflammatory bowel disease. *Gastroenterology*. 1994;106(2):287-296. https://doi.org/10.1016/0016-5085(94)90585-1

Irvine EJ, Zhou Q, Thomson AK. The short inflammatory bowel disease questionnaire: a quality of life instrument for community physicians managing inflammatory bowel disease. *Am J Gastroenterol.* 1996;91(8):1571-1578. https://doi.org/10.1186/s12955-021-01698-9

Kadel RP, Kip KE. A SAS Macro to Compute Effect Size (Cohen's) and its Confidence Interval from Raw Survey Data, SESUG2012

Mosli MH, Feagan BG, Zou G, Sandborn WJ, D'Haens G, Khanna R, Behling C, Kaplan K, Driman DK, Shackelton LM, Baker KA, MacDonald JK, Vandervoort MK, Samaan MA, Geboes K, Valasek MA, Pai R, Langner C, Riddell R, Harpaz N, Sewitch M, Peterson M, Stitt LW, Levesque BG. Reproducibility of histological assessments of disease activity in UC. Gut. 2015 Nov;64(11):1765-73. doi: 10.1136/gutjnl-2014-307536. Epub 2014 Oct 30. PMID: 25360036.

Reilly TJ, MacGillivray SA, Reid IC, Cameron IM. Psychometric properties of the 16-item Quick Inventory of Depressive Symptomatology: a systematic review and meta-analysis. *J Psychiatr Res.* 2015;60:132-140. https://doi.org/10.1016/j.jpsychires.2014.09.008

Rush AJ, Carmody T, Reimitz PE. The Inventory of Depressive Symptomatology (IDS): Clinician (IDS-C) and self-report (IDS-SR) ratings of depressive symptoms. *Int J Methods Psychiatric Res.* 2000;9:45-59. https://doi.org/10.1002/mpr.79

Spitzer RL, Kroenke K, Williams JB, Löwe B (May 2006). "A brief measure for assessing generalized anxiety disorder: the GAD-7". *Archives of Internal Medicine*. 166 (10): 1092–7. doi:10.1001/archinte.166.10.1092. PMID 16717171.

Steere, Boyd¹; Schmitz, Jochen¹; Powell, Nick²; Higgs, Richard¹; Gottlieb, Klaus¹; Liu, Yushi¹; Jia, Bochao¹; Tuttle, Jay L¹; Sandborn, William J³; Sands, Bruce E⁴; D'Haens, Geert⁵; Reinisch, Walter⁶; Krishnan, Venkatesh¹,\*. Mirikizumab regulates genes involved in ulcerative colitis disease activity and anti-TNF resistance: results from a phase 2 study. Clinical and Translational Gastroenterology ():10.14309/ctg.000000000000000578, March 07, 2023. | DOI: 10.14309/ctg.0000000000000578

Winthrop KL, Novosad SA, Baddley JW, et al. Opportunistic infections and biologic therapies in immune-mediated inflammatory diseases: consensus recommendations for infection reporting during clinical trials and postmarketing surveillance. Ann Rheum Dis. 2015;74(12):2107-2116. https://doi.org/10.1136/annrheumdis-2015-207841

Youden, W.J. Index for Rating Diagnostic Tests. Cancer. 1950; 3, 32-35.https://doi.org/10.1002/1097-0142(1950)3:1<32::AID-CNCR2820030106>3.0.CO;2-3